CLINICAL TRIAL: NCT04143880
Title: An International Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of Progesterone Combined Intranasal and Intramuscular Administration in Patients With Acute Hemorrhagic Stroke
Brief Title: Progesterone in the Treatment of Acute Hemorrhagic Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Korea University Anam Hospital (Other); Seoul National University Hospital (Other); Lishui Country People's Hospital (Other); Jinhua Central Hospital (Other); Huzhou Central Hospital (Other); The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YANWQ001
Record Dates: First submitted 2019-10-15; First posted 2019-10-29 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Progesterone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Progesterone
  Interventions: Drug: Progesterone
- control grou (Placebo Comparator): saline
  Interventions: Other: saline

INTERVENTIONS:
Drug: Progesterone — intramuscular injection intranasal administration
  Other Names: progesterone injection
  Arms: experimental group
Other: saline — intramuscular injection intranasal administration
  Arms: control grou

SUMMARY:
A large number of preclinical studies have confirmed that progesterone and its metabolites have strong neuroprotective effects. As a neuroprotective agent, progesterone has been effective in several animal models of nerve injury, suggesting that the drug has a wide range of neuroprotective effects. Pharmacodynamic studies have shown that some characteristic mechanisms of the action of the neurosteroid on brain injury and cerebral congestion include: prevention of inflammatory reaction and cell death (by inhibiting the activation of inflammatory cytokines and microglia); control of angiogenic brain edema (by reestablishing blood-brain barrier and regulating aquaporin-4 water transporter) and cytotoxic edema (by regulating Progesterone can also improve the neural dysfunction after cerebral hemorrhage, promote the regeneration and repair of damaged axons (activate PI3K / Akt pathway to inhibit the expression of RhoA), prevent the loss of Ca2 + caused by excitotoxicity and improve the survival rate of neurons. It was found that progesterone injection could reduce brain edema and promote the recovery of nerve function after brain injury.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to further evaluate the safety and effectiveness of progesterone in the clinical application of major cerebral congestion diseases. The Second Affiliated Hospital of Zhejiang University is the unit in charge of clinical research, and six units participate in the multicenter randomized, double-blind, placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute hemorrhagic stroke was confirmed by CT or MRI. There should be no obvious sequelae symptoms in the first stroke or previous stroke, Mrs < 2 (slight or no neurological dysfunction).
* Patients aged 40-80 (male, menopausal women);
* Patients with 6-48 hours of onset;
* 3 points ≤ NIHSS score ≤ 15 points for light and medium patients;
* Patients or family members sign informed consent.

Exclusion Criteria:

* Cerebral CT has excluded intracranial hemorrhage, and there is no imaging change of early large area cerebral infarction.
* Pregnant or lactating women;
* Previous intracranial hemorrhage, including suspected subarachnoid hemorrhage; large area stroke (> 2 / 3 MCA territory) or head CT showed any degree of midline displacement due to brain edema. Signs of intracranial hemorrhage (ICH, SAH, extradural hemorrhage, acute or chronic SDH) were found on baseline CT or MRI scan.
* Fever, defined as central body temperature > 37.5 ℃;
* Patients with severe heart, liver and kidney dysfunction or severe diabetes;
* Platelet count was less than 100 × 109 / L, blood glucose was less than 27 mmol / L, serum creatinine was more than 2.0 mg / dL or 180 μ mol / L.
* Blood pressure: systolic pressure > 180 mmHg, or diastolic pressure > 100 mmHg;
* Those who have previous allergic history to progesterone and citicoline;
* The anticoagulant has been taken orally, and INR is more than 15; heparin has been taken within 48 hours (APTT is beyond the normal range);
* Participating in clinical trials of any other treatment;
* Patients considered by the researchers not suitable for inclusion.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 3 month
  The percentage of patients with Mrs score 0, 1 and 2 was compared.